CLINICAL TRIAL: NCT02921191
Title: Descriptive Analysis of First-Cycle Prophylactic Use of G-CSF in Patients With Breast Cancer, Lung Cancer, or Lymphoma Treated With High Neutropenia Risk Chemotherapy
Brief Title: Descriptive Analysis of G-CSF Use in Patients With Breast Cancer, Lung Cancer, or Lymphoma Treated
Status: Completed | Type: Observational
Sponsor: Biologics & Biosimilars Collective Intelligence Consortium (Other)
Collaborators: Henry Ford Health System (Other); Aetna, Inc. (Industry); Amgen (Industry); College of Pharmacy, University of Nebraska College (Unknown); College of Pharmacy, University of New England (Unknown); HealthPartners Institute (Other); Momenta Pharmaceuticals, Inc. (Industry); Harvard Pilgrim Health Care (Other)
Responsible Party: Sponsor
Other Study IDs: BBCIC -GCFs
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Lung Cancer
Keywords: recombinant human granulocyte colony-stimulating factors; G-CSFs; biosimilar; biologics; High Neutropenia Risk Chemotherapy; Biologic and Biosimilars Collective Intelligence Consortium; bbcic
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms | interventions — Filgrastim; pegfilgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Lung cancer: Lung cancer patients receiving their first cycle of Grade III and IV myelosuppressive chemotherapy regimen treated prophylactically with G-CSF.
  Interventions: Drug: filgrastim, TBO-filgrastim or pegfilgrastim
- Breast cancer: Breast cancer patients receiving their first cycle of Grade III and IV myelosuppressive chemotherapy regimen treated prophylactically with G-CSF (filgrastim, TBO-filgrastim or pegfilgrastim)
  Interventions: Drug: filgrastim, TBO-filgrastim or pegfilgrastim

INTERVENTIONS:
Drug: filgrastim, TBO-filgrastim or pegfilgrastim — First cycle
  Other Names: Neupogen, Neulasta, Granix, Zarxio

SUMMARY:
Purpose:

With the existing recombinant human granulocyte colony-stimulating factors (G-CSFs) patents expiring and the FDA approval of new biosimilar and innovator biologics, patients being treated with Grade III and IV myelosuppressive chemotherapy regimens will have additional therapeutic options. This observational study will describe the patient characteristics of new users of G-CSFs. It will describe in the treatment cohorts a primary outcome of hospitalizations for febrile neutropenia. The BBCIC will use the findings from this descriptive analysis to design a comparative study evaluating the real-world effectiveness and safety of biosimilar and innovator G-CSFs.

DETAILED DESCRIPTION:
Additional information:

To most effectively interpret results from this descriptive analysis it is important to consider that this protocol was not designed to support a hypothesis. This information is being provided to the public in the interest of transparency and for demonstrating the BBCIC's Distributed Research Network's (DRN) ability to define exposures, outcomes, covariates and confounders. When published, the report will caution that the protocol does not support any ability to compare safety or effectiveness but instead is to be used only to explore the feasibility of future, more detailed comparative analyses and to better understand the capabilities of the BBCIC project. Further, the report will caution that information from this protocol should not affect use of the medical products described in any way and the fact that the BBCIC is performing this descriptive analysis in no way suggests there is a safety or effectiveness issue with any of the products described.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with baseline period of 183 days with continuous medical and pharmacy coverage preceding the first prescription fill for G-CSF
* Breast or lung cancer patients receiving their first cycle of Grade III and IV myelosuppressive chemotherapy regimen treated prophylactically with G-CSF.

Exclusion Criteria:

During baseline 365 days, any patient with a claim for (or with)

* Chemotherapy drug.
* Skilled nursing facility (SNF) or hospice care
* Diagnosis for a secondary breast cancer diagnosis
* A second cancer diagnosis (i.e., not breast, lung, lymphoma)
* Bone marrow or stem cell transplant
* Radiotherapy
* Chemo cycle >First: (exclude any chemotherapy cycles post the index G-CSF date)
* HIV/AIDS
* Hepatic disease
* Other non-oncology related neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects are selected according to inclusion criteria from a source population within the Sentinel Common Data Mode v5.0.1 (SCDM). The SCDM includes over 100 million individuals with 358 million person-years of observation time who are covered by Aetna, Anthem, Group Health Cooperative, Harvard Pilgrim Health Care, and HealthPartners. The time period assessed will be 1/1/2008-9/30/2015.
Sampling Method: Non-Probability Sample
Enrollment: 57725 (Actual)
Dates: Start 2008-01; Primary Completion 2015-09 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Hospitalizations for severe neutropenia | Anticipated completion February 2017
  Primary: Incidence of hospitalizations for febrile neutropenia in patients with breast or lung cancer receiving their first cycle of Grade III and IV myelosuppressive chemotherapy regimen treated prophylactically with G-CSF

SECONDARY OUTCOMES:
Incidence severe neutropenia | Anticipated completion February 2017
  Incidence severe neutropenia (ANC<0.5g/l)

CONTACTS AND LOCATIONS:
Overall Officials: Vanita Pindolia, PharmD, VP, Principal Investigator — Henry Ford Health Systems; Pam Pawloski, PharmD, Principal Investigator — HealthPartners Institute

IPD SHARING:
Plan to Share IPD: Yes
BBCIC Charter requires transparency and publication
Supporting Information: SAP
Time Frame: Publication is in press as of January 2021 in the Journal of the National Comprehensive Cancer Network. Pawlowski PM, McDermott CL, Marshall JH et al.
  "BBCIC Research Network Analysis of First-Cycle Prophylactic G-CSF Use in Patients Treated With High Neutropenia Risk Chemotherapy."

REFERENCES:
- [Background] AMCP Task Force on Biosimilar Collective Intelligence Systems; Baldziki M, Brown J, Chan H, Cheetham TC, Conn T, Daniel GW, Hendrickson M, Hilbrich L, Johnson A, Miller SB, Moore T, Motheral B, Priddy SA, Raebel MA, Randhawa G, Surratt P, Walraven C, White TJ, Bruns K, Carden MJ, Dragovich C, Eichelberger B, Rosato E, Sega T. Utilizing data consortia to monitor safety and effectiveness of biosimilars and their innovator products. J Manag Care Spec Pharm. 2015 Jan;21(1):23-34. doi: 10.18553/jmcp.2015.21.1.23. PMID 25562770
- [Background] Pawloski PA, McDermott CL, Marshall JH, Pindolia V, Lockhart CM, Panozzo CA, Brown JS, Eichelberger B. BBCIC Research Network Analysis of First-Cycle Prophylactic G-CSF Use in Patients Treated With High-Neutropenia Risk Chemotherapy. J Natl Compr Canc Netw. 2021 Aug 16:jnccn20268. doi: 10.6004/jnccn.2021.7027. Online ahead of print. PMID 34399406
- See also: The Biologics and Biosimilars Collective Intelligence Consortium (BBCIC) was established in 2015 to address anticipated needs for post-marketed evidence generation for novel biologics, their corresponding biosimilars and other related products. — http://bbcic.org